CLINICAL TRIAL: NCT01349062
Title: Phase III Clinical Studies on Traditional CAM Therapy in the Treatment of HIV/AIDS
Brief Title: Traditional Complementary and Alternative Medicine (CAM) Therapy in the Treatment of HIV/AIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Traditional Alternative Medicine Research, India (Other)
Responsible Party: Principal Investigator, RAMAKRISHNAN MADHUSOODANAN, Director, Traditional Alternative Medicine Research Center TAMRC-INDIA, Traditional Alternative Medicine Research, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00276991
Record Dates: First submitted 2011-05-03; First posted 2011-05-06 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: HIV Infections
Keywords: Prolonged Viral Suppression; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Immunotherapy

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "Kallunk oxide (Immunotherapy)" (Other): The participants will be received a daily regimen of "Kallunk oxide(Immunotherapy)" .
  Interventions: Drug: "Kallunk oxide (Immunotherapy) "

INTERVENTIONS:
Drug: "Kallunk oxide (Immunotherapy) " — The study is assigned Arm 1 above 450 cu/mm^3 baseline CD + T cells. HIV type-1 subjects will receive one drug, a daily regimen of "Kallunk oxide(Immunotherapy) + Long Pepper", that is a combination of a traditional alternative medicine (Complementary and Alternative Medicine CAM) as "Kallunk oxide" and appropriate drug carrier antidote. The drug assigns to 5 mg "Kallunk oxide" molecules with1995 mg "Antidote"( This antidote was used as a carrier of "Kallunk oxide" molecules), respectively, for children and adults. Dosage: 2000 mg for children and adults. This powder form sample size product will be administered once daily dose on 7 days treatment. The Botanical name of the antidote is "Piper Longum".
  Other Names: 'Kallide'

SUMMARY:
This research work is important for the cure/control of HIV infection. The study is intended to confirm the efficacy of "Kallunk Oxide (Immunotherapy)" molecules in the Treatment of HIV infection. The study will investigate the T- Lymphocytes (immune) response to HIV in order to boost the body's natural immune ability against infection. The basic study is directly inhibit a protein's increased functions, not only in the CD4+T cell but also CD3+ and CD8+ T cells and the CD45+. cells.

The 'Yogaprabhava', the drug's effectiveness, and progressive immunity with diet and lifestyle can be more easily studied.

DETAILED DESCRIPTION:
This research study is an individual investigator initiated meritorious project to confirm the efficacy of "Kallunk Oxide (Immunotherapy)" in the treatment of HIV- infection.The Previous clinical studies are showing that the T- Lymphocytes responses to "Kallunk Oxide (Immunotherapy)" is effective in the treatment of HIV- infection.

This randomized intervention study to confirm the efficacy of booster dose Kallunk Oxide molecules 5 mg to all participants,especially, greater than 8 years old children (Adolescence and Adults) , men and women. The Principal Investigator will be selected the informed consented patients to recruit for this trial. This study will be adhered by "Helsinki Declaration".

The patient's assays of Lymphocyte enumeration is the primary end point. Immune output of this drug and it's progressive immunity against HIV cure will follow- up. The study will be investigated the T- Lymphocytes (immune) response to HIV. The impact of the CD3+, CD4+,CD8 T cells and CD45+ response to "Kallunk Oxide (Immunotherapy)" will be studied.

Patient's body weight, CD4+ T cells and other hematological status will be investigated before and after the treatment period.

The research team is also mindful the symptoms such as nausea, fatigue and weight loss, sweating, shortness of breath, joint pain, etc. will individually being noted.

During this treatment period, in case, any of the patients have temperature, digestion complaint or chill, etc. may vary. Only in this circumstance,the patients not advised to use the controlled diet protocol or use of mutton soup, cow milk and cow ghee.

Privacy and Confidentiality:

The study must be handled a transparent privacy environment to recruit HIV-infected people all over India and the data will be confidentially protected with genuine written informed consent.

Dosage:

5 mg "Kallunk Oxide (Immunotherapy)" molecules with the antidote 1995 mg "Long Pepper"(Botanical name- Piper longum) for > 8 to < 45 years old children and adults from both genders.The study will also be evaluated the effectiveness of booster dose Kallunk Oxide (5 mg) and "Long Pepper" (1995 mg) in ART drug ( one tablet contains Zidovudine, lamivudine, and nevirapine ) using adults (<45) and adolescence (the ages12 to 18 years female and 14 to 18 years old male) to access serum negative status of HIV in CD+ T cell number <350 cu/mm^3 of ART using HIV-patients..

Favorable results on integrative intervention approach is point out that before using "Kallunk Oxide (Immunotherapy)' with ART is need nearly a six hour time frame. More meaningfully, it is stated that the HIV/AIDS patient may use ART at the evening time to avoid possible side effects as joint pain and fatigue (which are seldom cases).

The booster dose regimen of this therapy is administered as once daily dose for 10 days adherence for six months ART drug (Not Kallunk Oxide Therapy) tolerance. If the virus is not suppressed completely, drug resistance can develop. So, through this study the serum negative status of HIV from baseline to 24 weeks will be followed-up.

Dosage: powder form sample size product 2 gm (Kallunk Oxide + Antidote) for children and adults as once daily dose and is recommended to 7 days daily regimen for monthly use as mentioned baseline and six (6) months time frame.

Controlled Nourished diet:

Patients will be controlled by nourished diet protocol. Eat wheat products, rice food products, cow milk (only ½ cup), cow ghee, green gram,banana, mutton soup,sweet fruits as apple (only sweet), orange and prepared black pepper added vegetable foods.

Restriction:

Salts, other oils, mustard,Pumpkin,lemon juice, and tamarind fish items are not use within 10 days of medication.

Drug Administration:

In this study, patients can use the capsule/powder form medicine with 1/2 cup hotter water. HIV- patients be used one drug "Kallunk oxide (Immunotherapy)" as calcined/or oxidized molecules.

Precaution:

No precaution is needed. The patients can avoid sediments at the bottom of the cup.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HIV/AIDS
* Able to swallow tablets or powder form medicine
* Able to eat nutritional foods
* HIV infected patients
* Signed consent of parent or guardian for patients under 18 years of age
* Interest to use of study drugs
* Follow at a participating clinical site and
* Children greater than 8 years old.

Exclusion Criteria:

* Medical side effects
* Pregnant or breast feedings
* History of significant cardiac abnormalities or dysfunction
* Received certain drugs (Steroid) or treatments
* Unable to followed at a participating clinical center
* Children less than 8 years old
* Any serious conditions (severe chronic stage AIDS cases) at study entry that may affect the results of the study.
* Allergy to any of the study drugs or their formulations
* Tobacco using patients
* Alcohol using patients and
* Drug addicting patients.

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Actual)
Dates: Start 2012-02-27 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Efficacy | Number of Participants with Adverse Events by weeks 24
  Number of participants with adverse events for efficacy by mentioned time frame will be assessed.

SECONDARY OUTCOMES:
Viral Load Assay | Three months follow up
Absolute Immune Cells Count Assay(CD3, CD4, and CD8 + T cells) | Three months follow up study
Prolonged Viral Suppression | Six Month's Follow up study

CONTACTS AND LOCATIONS:
Overall Officials: Ramakrishnan Madhusoodanan, PHD, Principal Investigator — Traditional Alternative Medicine Research Center
Locations (3):
- India (3):
  - Project Site Office, Near Sivan Kovil, Nallepily, Hospital of Integrated Research Site HIRS [new]), Palakkad, Kerala
  - Project Site Office, Hospital of Integrated Research Site HIRS(New), Karoor, Ambalapuzha-PO, Alleppey-District, Kerala, India 688561, Alappuzha
  - Project Site Office, Hospital of Integrated Research Site HIRS(New), Ahammed Nagar, Mathura Nagar, Bhingar- PO, Mumbai

IPD SHARING:
Plan to Share IPD: No